CLINICAL TRIAL: NCT03210636
Title: Feasibility and Safety Study of LapSpace, A Novel Laparoscopic Surgical Instrument
Brief Title: Looking at Safety and Feasibility of Novel Laparoscopic Device (LapSpace)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: LapSpace Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00035940
Record Dates: First submitted 2014-10-23; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Patients Undergoing Laparoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- With Use of LapSpace (Experimental): evaluate ease of use, safety evaluations, surgeon and clinician feedback
  Interventions: Device: LapSpace

INTERVENTIONS:
Device: LapSpace — use of atraumatic laparoscopic retractor for patients undergoing laparoscopic surgery

SUMMARY:
In order to help the surgeons to clearly visualize their target operating area and create an optimal operative field throughout the procedure, the device owners have developed a new class of inflatable laparoscopic retractors for both bowel and organ specific retraction with load bearing bore by an inflatable reinforced material that is atraumatic, biocompatible, and are self-retained, i.e. require no personnel to maintain them post-placement.

Specifically, the device owners menu of designs hold a range of 50 - 100 % of the bowels and support at minimum 6 lbs in the vertical direction. All the device owners devices enter the abdominal cavity through a conventional 10mm incision. The pressure within the inflatable tubes of the device will not be above 15 mmHg, which is the current pressure used to insufflate the patient's abdomen with carbon dioxide (CO2). The devices are able to retract up to 10 cm of the bowels in any direction within the coronal plane and retract the bowels 10cm upward, towards the abdominal wall. Finally, the invention here-in described can be manipulated easily to provide retraction of specific organs, including, liver, bladder, uterus, etc.

The device has been approved by the FDA for clinical use (FDA Registered) and the purpose of this study is to evaluate the device in laparoscopic operations for safety and feasibility.

DETAILED DESCRIPTION:
The field of laparoscopy has been growing exponentially during the past decade because of its tremendous benefits over open surgery such as minimal incisions, lesser post-operative trauma, quicker recovery, lesser scarring, reduced hospital stay and lower infection rates. It is clear that the success of any laparoscopic surgery lies on the optimal exposure of the operative site. Surgeons and assistants are required to tightly strap the patients on the surgical bed, continuously change the patient's position in order to use gravity to hold the bowels out of the way and finally result in manual over manipulation of bowels and organs using graspers in order to achieve the optimal exposure of their site. However, small bowels or organs cannot be held back efficiently using these techniques and slide continuously into the operating area.

In practice, the obstruction of the surgeons' visual field and the excessive manipulation of the bowels cause unintentional injuries, bleeding, bruising, hematoma and perforations that might require patients to undergo

additional surgeries because of scar tissue formation. The U.S market for scar tissue prevention products is estimated at a staggering $2-3 billion. Furthermore, the current standard of clinical care forces surgeons to add procedural steps in the operation in order to minimize possible complications. However, these extra steps further extend the duration of the operations, leading to a loss of money and reliability on behalf of the hospitals.

The device owners bowel retractors eliminate the time-consuming mobilization of the small intestines while they stabilize the bowels, allowing for a clear view of the operative site. Given the increased demand of laparoscopic surgeries in which the device owners device is helpful (approaching 5 million surgeries per year) the time saved after only a few uses of the device owners device is significant enough to benefit hospitals in allowing them to host another surgery that is waiting in the backlog. The device owners devices, thus, are not only beneficial for the patients since they minimize trauma and complications but also highly profitable for the hospitals.

The proposed device contains a variety of novel features, which are enumerated henceforth. The device owners device will be inflatable and will have inflatable "ribs" at the grasping terminal of the device. The ribs will work in tandem with the mechanism of inflation in order to adequately grasp the desired portion of bowel in the abdominal cavity. In addition, the device owners device will be firmly attached to a solid steel center rod, with which the surgeon can maneuver the device. The solid rod will also contain a sliding seal, such that after the device has been inserted into the abdominal cavity, the seal can be slid into place and will serve to effectively anchor the device on the abdominal wall. On the end of the rod near the surgeon, there will be an attached handle with a trigger. This handle system will be used to inflate the device by pulling the trigger and allowing compressed air through the central rod. The handle will also be the point of contact between the surgeon's hand and the device owners device, allowing him further maneuverability throughout the procedure.

The product is a bowl-shaped device that is intended to be used as an organ or bowel retractor in laparoscopic surgeries. This device consists of a central, hollow rod made of steel that has a straight proximal end and a curved distal end. The aforementioned distal end of the device has an inflatable portion, the material for which encircles the central rod. The inflatable portion also contains tubular projections which emanate from where the material contacts the central rod out to the edges of the inflatable portion. These projections are denoted henceforth as "ribs". The inflatable material is a biocompatible polymer that can hold sufficient tension and pressure for the application of laparoscopic surgery. The ribs curve inwards, which create a bowl-like structure when fully inflated and deployed. Each of the ribs are connected to the central rod and to each adjacent rib via membrane, which is connected medially to the central shaft all along the distal, curved end. This creates a functional inflatable endoskeleton to support the bowels and organs that will be in contact with this device during laparoscopic surgery. The amount of inflation of the device can be modulated by the surgeon, by increasing or decreasing the inflation pressure as desired by adding more compressed air or withdrawing compressed air, respectively.

The proximal end of the central rod will have a handle grip with a trigger attached to it. There will be an inlet for where a canister of compressed air will be positioned, such that when the trigger is depressed by the surgeon, air will flow down the length of the hollow central rod and inflate the device. The handle and grip

will be attached such that the surgeon can deftly maneuver and retract the device after it has been inserted in the patient.

The central rod will further house a sealing mechanism that can slide along the length of the rod, from the proximal handle to the distal end. This sliding seal will be affixed in place to the abdominal wall, allowing for a functional anchor and pivot point about which the retractor has many degrees of freedom with respect to movement, while still being supported by the seal to the patient's abdomen. A surgeon can choose to use a trocar in lieu of a sliding seal, which will have to be placed on the central before the attachment of the handle grip.

After the device is in place after being fully inflated, it has the ability to grasp and hold the bowel in its concave interior region. The ribs help maintain the accurate shape and rigidity of the inflated portion, and thus will allow the device to remain flush against the bowel during retraction. The surgeon will then

presumably pull the central rod to a more beneficial location, such that the operative field is no longer obstructed by the device. The surgeon can then affix the device to a surgical bed clamp, so as to free the surgeon from holding the device in place throughout the duration of the procedure.

As of now, the device is to be utilized for laparoscopic abdominal surgical procedures. However, a similar or slightly modified product could be used for gynecological procedures as well, and would aid in the retraction or holding of pelvic or lower abdominal organs in those procedures. In addition, future variations of the design could be applicable to upper abdominal or cardiothoracic procedures as well. This device could also potentially be used in organ resection as well as retraction, in that modifications to the device could potentially allow it to clear the operative field while simultaneously being involved in organ excision.

ELIGIBILITY:
Inclusion Criteria:

* consenting adults between the ages of 18 to 65
* patients undergoing laparoscopic operations
* english-speaking patients
* patients who are capable of consenting for their own operation
* non-emergent, elective cases

Exclusion Criteria:

* non-laparoscopic cases
* emergent cases
* no witnessed consent
* children and elderly adults age >65
* non-english speaking patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Surgeon preference | immediately following surgery, up to 2 hours
  surgeon questionnaire given to measure preference using a rating of 1 to 5 with 1 being "would not use to 5 being "I would use"